CLINICAL TRIAL: NCT04746170
Title: The Effect of Labor Dance Applied to Pregnant Women in the First Stage of Labor on Labor Pain, Anxiety, Birth Time and Maternal Satisfaction at Birth: A Randomized Controlled Study
Brief Title: The Effect of Labor Dance on Labor Pain, Anxiety, Birth Time and Maternal Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Dilek Kaloglu Binici, Research Assistant, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Labor Dance
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pregnant Women
Keywords: Birth; Labor Dance; Anxiety; Maternal Satisfaction; Nurse
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study was planned as a randomized controlled trial. The pregnant will be followed in single rooms. Pregnant women in the experimental group will be given labor dance with music for 15 minutes per hour until the cervical opening starts from 3 cm (latent phase) and the cervical opening reaches 8 cm.
Who Masked: Participant, Outcomes Assessor
Masking Description: In RCT, blinding will be done in terms of participants and statistics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multiparous (Experimental): Pregnant women in the experimental group will be given a labor dance with music for 15 minutes per hour until the cervical opening starts from 3 cm (latent phase) and the cervical opening reaches 8 cm. The massage application will be made by the researcher to their waist and sacrum area with a ball massage glove.
  Interventions: Other: Labor Dance
- Multiparous Control (No Intervention): Only routine practices were performed with the control group, and data were recorded as in the experimental groups.
- Primipar (Experimental): Pregnant women in the experimental group will be given a labor dance with music for 15 minutes per hour until the cervical opening starts from 3 cm (latent phase) and the cervical opening reaches 8 cm. The massage application will be made by the researcher to their waist and sacrum area with a ball massage glove.
  Interventions: Other: Labor Dance
- Primiparous control (No Intervention): Only routine practices were performed with the control group, and data were recorded as in the experimental groups.

INTERVENTIONS:
Other: Labor Dance — Pregnant women in the experimental group will be given a birth dance with music for 15 minutes per hour until the cervical opening starts from 3 cm (latent phase) and the cervical opening reaches 8 cm. The massage application will be made by the researcher to their waist and sacrum area with a ball massage glove.
  Arms: Multiparous; Primipar

SUMMARY:
Pregnant women who are in the process of labor need physical and emotional support of health professionals in issues such as coping with labor pain, relieving fear and anxiety, and experiencing positive birth. The fact that labor dance includes components such as upright posture, pelvic movement, touch, massage provides both physical and emotional support to the pregnant woman. The aim of the study is to examine the effect of labor dance applied to pregnant women in the first stage of birth on labor pain, anxiety, birth time and maternal satisfaction at birth.

DETAILED DESCRIPTION:
The study was planned in randomized controlled experimental type. The pregnant women will be followed in single rooms. The information about how to apply the labor dance to the pregnant women in the experimental group will be explained by the researcher in the latent phase of birth and will be shown practically. Pregnant women in the experimental group will be given labor dance with music every hour until the cervical opening starts from 3 cm (latent phase) and the cervical opening reaches 8 cm. Pregnant women will musically choose one of Acemaşiran Authority, Rehavi Authority and Farid Farjad's Thin Rose of My Idea. The researcher and pregnant women will perform a labor dance with the music for 15 minutes per hour. The researcher and the pregnant will hold each other's hands (3-4 steps distance), stand opposite each other and perform pelvic tilt together. When the pregnant woman desires or has contractions, the researcher will massage the waist and sacrum area with a ball massage glove.

Details of the application and birth (such as dance time, birth time, contractions) will be recorded by the researcher. Pregnant women will be followed by the doctor, midwife and researcher during the tram, birth and first four hours postpartum.

Ball Massage Glove Used in Mechanical Massage Application It consists of nine metal balls with a diameter of 1.5 cm that can rotate 360 degrees. With its glove design and ergonomic structure, it can be easily applied to any area. By concentrating directly on the massage points, it can be used more effectively on all points of the body. Since it is made of silicone material, it does not harm the hand and the area to be massaged while massaging. (Information taken from introductory guide).

ELIGIBILITY:
Inclusion Criteria:

* Not being pregnant diagnosed with Covid -19 (last 20 days)
* Accepting to be included in research,
* 20 years of age,
* Speak Turkish,
* At least a primary school graduate,
* No disability such as hearing or vision,
* Having a pregnancy at term (those between 38-41 weeks of gestation),
* Pregnant women whose labor has started actively,
* Applying to the delivery room for vaginal delivery in the latent phase of labor (when the cervical opening is 1-3 cm),
* Pregnant women without uterine contraction anomaly,
* Having a single fetus, The leading part of the fetus is the head coming (in the vertex position),
* Fetus weight 2500-4000 gr,
* Being in the low risk pregnant group (Absence of conditions such as placenta previa, preeclampsia, heart, gestational diabetes, intrauterine growth retardation, intrauterine dead fetus, macrosomic babies, fetal distress etc.),

Exclusion Criteria:

* Pregnant women whose previous birth type was cesarean section (pregnant women who preferred vaginal delivery after cesarean section)
* Pregnant women who received epidural analgesia,
* Pregnant women whose labor lasted less than 3 hours (rapid birth story).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | During labor assessed up to 12 hours
  VAS is used to measure perceived pain. The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on lower end (no pain) and on upper end (extreme pain). The pregnant women is asked to mark their current pain level on the line.
State Anxiety Scale | During labor assessed up to 7 hours
  The scale consists of 20 items. The emotions or behaviors expressed in the articles are according to the degree of feeling the situation in which the individual is; It is answered by marking one of the options such as (1) none, (2) a little, (3) much, (4) completely. The total score obtained from the scale is between a minimum of 20 and a maximum of 80. The last value obtained is the individual's anxiety score.
State Anxiety Scale | within the first 4 hours postpartum
  The scale consists of 20 items. The emotions or behaviors expressed in the articles are according to the degree of feeling the situation in which the individual is; It is answered by marking one of the options such as (1) none, (2) a little, (3) much, (4) completely. The total score obtained from the scale is between a minimum of 20 and a maximum of 80. The last value obtained is the individual's anxiety score.

SECONDARY OUTCOMES:
The Scale for Measuring Maternal Satisfaction (SMMS)-normal birth | within the first 4 hours postpartum
  The scale consists of 43 and 10 sub-dimensions. The sub dimensions of the scale; perception of the healthcare team, midwifery-nursing care in labor, relief, participation in decisions and information, respect for privacy, meeting expectations, meeting the baby, postpartum care, hospital room and hospital facilities. The items of the scale are scored on a 5-point Likert-type scale according to whether they agree with the statements or not. The answers given by the items (1-2-3-4-5 / Disagree-Partially Agree-Undecided-Agree-Strongly Agree) are scored on a five-point Likert-type scale depending on whether the items agree with the statements or not. The total raw score is the lowest 43 and the highest 215. As the total score obtained from the scale increases, the level of satisfaction of mothers with the care they receive in the hospital during normal delivery increases.
Labor duration was assessed with The Postpartum Maternal Information Form (PMIF) | During labor assessed up to 18 hours
  The Postpartum Maternal Information Form (PMIF) was prepared by the researchers using the relevant literature. It consists of questions regarding information about birth (duration of labor, oxytocin, and episotomy practices at birth)

CONTACTS AND LOCATIONS:
Overall Officials: Dilek KALOĞLU BİNİCİ, Principal Investigator — Artvin Coruh University
Locations (1):
- Artvin State Hospital, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akin B, Saydam BK. The effect of labor dance on perceived labor pain, birth satisfaction, and neonatal outcomes. Explore (NY). 2020 Sep-Oct;16(5):310-317. doi: 10.1016/j.explore.2020.05.017. Epub 2020 May 30. PMID 32527687
- [Derived] Kalog Lu Binici D, Aktas S. The Effect of Labor Dance in the First Stage of Labor on Labor Pain, Anxiety, Duration of Labor, and Maternal Satisfaction with Labor: A Randomized Controlled Study. J Integr Complement Med. 2024 Apr;30(4):383-393. doi: 10.1089/jicm.2022.0818. Epub 2023 Oct 13. PMID 37831917